CLINICAL TRIAL: NCT02670291
Title: Treatment of Auditory Hallucinations in Schizophrenia With Bilateral Theta Burst Stimulation
Acronym: cTBS-AH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: German Research Foundation (Other); Institute for Clinical Epidemiology and Applied Biometry, University Tuebingen, Germany (Unknown); Center for Clinical Studies, University Tuebingen (ZKS), Germany (Unknown); Department of Psychiatry and Psychotherapy, University Munich (LMU), Germany (Unknown); University of Ulm (Other); Department of Psychiatry and Psychotherapy; University Heidelberg, Germany (Unknown); Department of Psychiatry and Psychotherapy; Unversity Augsburg, Germany (Unknown); Department of Psychiatry and Psychotherapy, LVR Duesseldorf, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PL 525/4-1
Record Dates: First submitted 2016-01-26; First posted 2016-02-01 (Estimated); Last update posted 2024-03-25 (Actual); Status verified 2022-06

CONDITIONS: Auditory Hallucinations; Schizophrenia
Keywords: auditory hallucinations; schizophrenia; cTBS; noninvasive brain stimulation
MeSH Terms: conditions — Hallucinations; Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- active cTBS (Active Comparator): Determination of resting motor threshold (RMT); Coil position: temporoparietal cortices halfway between T3/P3 and T4/P4 (EEG 10/20 system); active cTBS (80% of RMT);
  Interventions: Device: MagPro Cool-B65A/P, Magventure
- Sham cTBS (Sham Comparator): Determination of resting motor threshold (RMT); Coil position: temporoparietal cortices halfway between T3/P3 and T4/P4 (EEG 10/20 system); sham cTBS;
  Interventions: Device: MagPro Cool-B65A/P, Magventure

INTERVENTIONS:
Device: MagPro Cool-B65A/P, Magventure — combined active and sham coil
  Arms: active cTBS
Device: MagPro Cool-B65A/P, Magventure — combined active and sham coil
  Arms: Sham cTBS

SUMMARY:
This randomized, sham-controlled, double blind, multicentre clinical trial aims at providing evidence for the efficacy and safety of continuous theta burst stimulation (cTBS) in the treatment of auditory hallucinations in patients with schizophrenia. Overall, the study will include 137 patients. Because of the adaptive study design, an interim analysis was performed after half of the originally planned patients (43/86), according to which the sample size was increased by 51 patients). Each patient will receive a three weeks course of daily (5/week) treatment; 50% of the patients will be treated with cTBS (1200 impulses daily), the other half with a sham stimulation to the left and right temporoparietal cortex. Sham stimulation will be applied by an active sham-coil that allows for a double-blind treatment. Follow-up assessments 1, 3 and 6 months after treatment will investigate the stability of treatment effects.

DETAILED DESCRIPTION:
Auditory verbal hallucinations (AH), a cardinal feature of schizophrenia, are often severely distressing and increase the risk for violence and suicide. Although antipsychotic medication mostly exerts rapid beneficial effects on this symptom particularly in first-episode patients who continue on taking their medication (Sommer et al. 2012), in up to 25%-30% of all patients, such hallucinations persist (Shergill et al. 1998). The often progressive course of the disease and insufficient treatment adherence due to unwanted side effects significantly limit the treatment response. In turn, this lack of treatment efficacy also contributes to low treatment adherence which is generally associated with an unfavorable course of schizophrenia and increased relapse and readmission rate. New and effective treatments are therefore essential to reduce the massive individual burden and psychosocial costs associated with schizophrenia. Nevertheless, in the last decades, the hopes for new pharmacological treatment options have been disappointed and the pharmaceutical industry has apparently withdrawn from the development of new compounds for this disorder. Accordingly, the development of non-pharmacological approaches based on an increasing body of patho-physiological knowledge is even more needed to pave new ways for the treatment of this frequently detrimental symptom of schizophrenia.

The main objective of the present study is to provide high-level evidence for efficacy and safety of continuous theta burst stimulation (cTBS) in the treatment of auditory hallucination (AH) by this first full-size multicenter (3 centers) controlled clinical trial.

This is a double blind (actually triple blind, i.e. patient, clinical investigator, and person who will administer cTBS), randomized, sham-controlled clinical trial to test the efficacy and safety of bilateral (successively applied) daily cTBS to the temporoparietal cortex on the severity of AH. The study will be conducted in a two-armed parallel design in which 50 % of the patients will be treated with the verum stimulation and the other half of patients will receive the placebo / sham stimulation.

The cTBS protocol follows the method by Huang et al. (2005) and our pilot study (Plewnia et al. 2014a) to achieve a lasting reduction of cortical excitability. Accordingly, each stimulation train (40 s) of cTBS consists of 600 stimuli applied in bursts of 3 pulses at 50 Hz given every 200 ms (5 Hz). Stimulation intensity is standardized at 80% of the resting motor threshold (RMT) and applied successively to each hemisphere. For the first session, the order of right and left hemisphere will be determined by randomization and will alternate in each following session to preclude order effects.The RMT will be determined using EMG recordings from the left and right abductor pollicis brevis and defined as the minimal stimulation intensity needed to elicit at least 10 out of 20 motor-evoked-potentials of ≥ 50µV. RMT will be determined once, i.e. before the beginning of treatment period. The cTBS or sham treatment will be targeted both temporoparietal cortices halfway between T3/P3 and T4/P4 (EEG 10/20 system).

The treatment (active cTBS or sham cTBS) will be administered over a period of 3 consecutive weeks at each workday (Monday to Friday), resulting in a total of 15 treatment sessions. Ratings will be performed after the last treatment of each week by an independent rater. Follow-up visits are planned 1, 3 and 6 months after end of treatment phase to control for sustainability of cTBS treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age 18-65 years
* Schizophrenia (DSM-5 295.90), schizophreniform disorder (DSM-5, 295.40), or schizoaffective disorder (DSM-5 295.70)
* Auditory hallucinations (AH) present at least once a week, for at least 3 months
* No sufficient effect of at least one adequate antipsychotic treatment
* Severity according to PANSS hallucination score (Item P3) of 3 or more
* Fluent German language
* Stable antipsychotic medication 2 weeks before and 3 weeks during the treatment

Exclusion Criteria:

* Suicidality
* History/evidence of brain surgery
* Significant brain malformation or neoplasm
* Head injury
* Cerebral vascular events
* Neurodegenerative disorder
* Deep brain stimulation
* Intracranial metallic particles
* History of seizures
* Diagnose of substance dependence or abuse as primary clinical problem
* Severe somatic comorbidity
* Cardiac pacemakers
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2023-11 (Actual); Study Completion 2024-03 (Actual)

PRIMARY OUTCOMES:
Change of Psychotic Symptom Rating Scales - Auditory Hallucinations subscale (PSYRATS-AH) | 3 weeks
  Group comparison (active vs. sham cTBS) regarding the change of the auditory hallucination subscale of the Psychotic Symptom Rating Scales (PSYRATS-AH) score from baseline to end of treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Plewnia, Prof. MD., Principal Investigator — Dept. Psychiatry and Psychotherapy, Universtiy of Tuebingen
Locations (1):
- Department of Psychiatry and Psychotherapy, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Plewnia C, Brendel B, Schwippel T, Becker-Sadzio J, Hajiyev I, Pross B, Strube W, Hasan A, Campana M, Padberg F, Mayer P, Kujovic M, Lorenz S, Schonfeldt-Lecuona C, Otte ML, Wolf RC, Hoppner-Buchmann J, Serna-Higuita LM, Martus P, Fallgatter AJ. Theta burst stimulation of temporo-parietal cortex regions for the treatment of persistent auditory hallucinations: a multicentre, randomised, sham-controlled, triple-blind phase 3 trial in Germany. Lancet Psychiatry. 2025 Sep;12(9):638-649. doi: 10.1016/S2215-0366(25)00202-0. Epub 2025 Aug 4. PMID 40774272
- [Derived] Plewnia C, Brendel B, Schwippel T, Martus P, Cordes J, Hasan A, Fallgatter AJ. Treatment of auditory hallucinations with bilateral theta burst stimulation (cTBS): protocol of a randomized, double-blind, placebo-controlled, multicenter trial. Eur Arch Psychiatry Clin Neurosci. 2018 Oct;268(7):663-673. doi: 10.1007/s00406-017-0861-3. Epub 2017 Dec 9. PMID 29224040